CLINICAL TRIAL: NCT02599805
Title: Can Topical Oxygen Therapy (Natrox™) Improve Wound Healing in Diabetic Foot Ulcers?
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: tba
Record Dates: First submitted 2015-08-13; First posted 2015-11-09 (Estimated); Last update posted 2015-11-09 (Estimated); Status verified 2015-11

CONDITIONS: Diabetic Foot
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Natrox treatment group (Experimental): In this group, all subjects will have the Natrox™ ODS will be applied to the ulcer and attached to the active Natrox™ Oxygen Generator using the tubing provided or regular dressing will be used. Dressings according to the standard practice guidelines will be used. Patients in this group will continue to receive treatment as described by the diabetic foot ulcer standard of care. The ulcer will be photographed at biweekly intervals for a period of 8 weeks to analyze ulcer surface area using a standardized digital imaging software.
  Interventions: Device: Natrox™ Oxygen Delivery System (ODS)
- Control group (No Intervention): All subjects in this group will receive the Diabetic foot ulcer standards of care which include:
  * Full medical assessment in all cases.
  * Surgical operation/Intervention where indicated.
  * Local treatment of the ulcer (debridement followed by ulcer care according to "modern ulcer healing" standards and management of diabetes.) The ulcer will be photographed at biweekly intervals for a period of 8 weeks to analyze ulcer surface area using a standardized digital imaging software.

INTERVENTIONS:
Device: Natrox™ Oxygen Delivery System (ODS) — Natrox™ ODS will be applied to the subject's diabetic ulcer and attached to the active Natrox™ Oxygen Generator using the tubing provided or regular dressing will be used. The Natrox™ oxygen delivery system (ODS) is a device designed to overcome a number of problems associated with previous methods of oxygen therapy by delivering continuous oxygen to the ulcer bed through a dressing.
  Arms: Natrox treatment group

SUMMARY:
Diabetic foot complications care represent a significant burden to the Canadian healthcare system. The estimated annual expenditure in Canada for diabetic foot ulcers is more than $150 million. A small sized randomized controlled trial (n=17) investigating the use of topical oxygen therapy (n=9) against placebo (n=8) for diabetic ulcers was done recently and showed a 87% average reduction of ulcer size in treatment group versus 46% average reduction in the control group (p<0.05).

Despite the standards of care used today in diabetic foot ulcer treatment, wounds may be non-healing when they do not heal within the appropriate time frame expected by an experienced clinician. Current diabetic foot ulcer standards of care include: full medical assessment in all cases, surgical intervention where indicated and local treatment of the ulcer.

Given the scarcity of controlled trials specifically designed to review the effects of topical oxygen in ulcer care, this study will contribute to the understanding of the management of these ulcers by assessing the reductions in ulcer size achieved using Natrox™ topical oxygen therapy.

DETAILED DESCRIPTION:
Diabetic foot complications care represent a significant burden to the Canadian healthcare system. The estimated annual expenditure in Canada for diabetic foot ulcers is more than $150 million. Topical oxygen therapy has historically been recognized as essential for its antibiotic properties and as a nutrient. A number of studies have suggested that this method of treatment may contribute to better healing of wounds, particularly in ulcers. The Natrox™ oxygen delivery system (ODS) is a device designed to overcome a number of problems associated with previous methods of oxygen therapy by delivering continuous oxygen to the ulcer bed through a dressing. It consists of a small battery-powered oxygen concentrator which processes oxygen from air, is portable, and can be held in place by a lightweight strap. In this study, we will seek to determine the effectiveness of the Natrox™ Topical Oxygen device in patients with non-healing diabetic foot/leg ulceration in conjunction with standard best practice. The Diabetic foot ulcer standards of care include:

* Full medical assessment in all cases.
* Surgical operation/Intervention where indicated.
* Local treatment of the ulcer (debridement followed by ulcer care according to "modern ulcer healing" standards and management of diabetes.)

In both the treatment group and the control group, comparative changes in ulcer surface area will be measured over a period of 8 weeks to analyze wound healing.

ELIGIBILITY:
Inclusion Criteria

1. Diabetic foot ulcer, which has had optimum multi-disciplinary team management for >4 weeks
2. No planned treatment to arterial disease
3. No planned surgical intervention
4. Patients aged >18 years.
5. Patients who understand the study, agree to adhere to the treatment and are able to give consent
6. Patients who can be followed by the same investigating team for the whole period of their participation in the study

Exclusion Criteria

1. Presence of invasive infection requiring intravenous antibiotics
2. Presence of Methicillin-resistant Staphylococcus aureus (MRSA) or Pseudomonas aureus in the swab cultures
3. Pure Neuropathic ulcer with no arterial insufficiency unless they fail to heal within 12 weeks of optimum management
4. Significant reduced immunity or high dose corticosteroids (>10mg Prednisolone) or other second line immune-suppressant
5. Need for total contact cast
6. Patients with a known sensitivity to any of the components of the evaluation device
7. Patients with known or suspected malignancy in the ulcer or surrounding tissue.
8. Patients who do not have the physical or mental capacity, or a significant other with the ability to change the Natrox™ battery pack on a daily basis
9. Patients who present with more than 10% of the ulcer surface area covered in hard eschar
10. Patients with ulcer surface area of more than 10x10cm
11. Patients who are participating in another clinical study for ulcer management
12. Patients with a known history of poor compliance with medical treatment
13. Patients who are unable to understand the aims of the study and not give informed consent
14. Pregnant female patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Comparative change in ulcer surface area | 8 weeks
  Comparative change in ulcer surface area in the study group undergoing treatment with the NatroxTM ODS (n=10) after the 8 week treatment period. These changes in ulcer surface area will be compared to the changes measured in the control study group.

REFERENCES:
- [Background] Public Health Agency of Canada. Unpublished analysis using 2000 data from the Economic Burden of Illness in Canada. (Public Health Agency of Canada); 2009.
- [Background] Mani R (2010) Topical oxygen therapy for chronic wounds: a report on the potential of Inotec® a new device for delivering enriched oxygen to chronic wounds
- [Background] Driver VR, Yao M, Kantarci A, Gu G, Park N, Hasturk H. A prospective, randomized clinical study evaluating the effect of transdermal continuous oxygen therapy on biological processes and foot ulcer healing in persons with diabetes mellitus. Ostomy Wound Manage. 2013 Nov;59(11):19-26. PMID 24201169